CLINICAL TRIAL: NCT01612494
Title: Hypertonic Saline as Therapy for Pediatric Concussion: A Randomized Controlled Trial in the Emergency Department
Brief Title: Hypertonic Saline as Therapy for Pediatric Concussion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Angela Lumba, MD, Fellow, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HTS-100423
Record Dates: First submitted 2012-05-29; First posted 2012-06-05 (Estimated); Results first posted 2014-03-21 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Saline Solution, Hypertonic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal Saline (Placebo Comparator)
  Interventions: Other: Normal Saline
- Hypertonic Saline (Experimental)
  Interventions: Drug: Hypertonic Saline

INTERVENTIONS:
Drug: Hypertonic Saline — intravenous formulation of 3% hypertonic saline in a bolus dose of 10ml/kg over one hour
  Other Names: 3%; HTS
  Arms: Hypertonic Saline
Other: Normal Saline — intravenous formulation of normal saline in a bolus dose of 10ml/kg over one hour
  Other Names: NS
  Arms: Normal Saline

SUMMARY:
This single center, blinded, randomized controlled trial evaluated the use of hypertonic saline versus normal saline as therapy for the symptoms of pediatric concussion post head injury.

The study hypothesis was that hypertonic saline would improve symptoms of pediatric concussion following head injury as measured on the self-reported Wong Baker Faces Pain Scale as compared to normal saline.

The null hypothesis was that there would be no difference in change of reported pain in either group.

ELIGIBILITY:
Inclusion Criteria:

* 4-17 years old
* consent obtained
* pain as a symptom of concussion
* head CT negative for intracranial pathology

Exclusion Criteria:

* younger than 4 years or older than 17 years
* multi trauma
* cardiac, neuro, renal history of disease
* seizure
* narcotic, drug use
* pregnancy
* head CT with traumatic intracranial pathology
* no consent

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2010-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela K Lumba, MD, Principal Investigator — University of California, San Diego; Mary Hilfiker, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Rady Children's Hospital Emergency Department, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited over the course of one year from a single center's pediatric emergency department
Pre-assignment Details: No enrolled patients were excluded from the trial
Period: Overall Study
Arm/Group | Normal Saline | Hypertonic Saline
Started | 21 | 23
Completed | 21 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Hypertonic Saline | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 23 | 44
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.9 (3) | 12.1 (2.5) | 12 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 11 | 17 | 28
Region of Enrollment [Number; unit: participants]
  United States | 21 | 23 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain
Description: Self-reported pain assessment using the Wong-Baker Faces Pain Rating Scale. There are 6 faces with 5 intervals. Faces are numbered 0 to 10. Maximum score is the 6th face/10. Minimum score is the first face/0. Increasing faces represent increase in pain, decreasing faces represent decrease in pain. No subscales were included.
Time Frame: Following therapy to 2-3 days post discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Normal Saline | Hypertonic Saline
Number analyzed (Participants) | 21 | 23
units on a scale | 1.14 (1.5) | 3.5 (1.6)

ADVERSE EVENTS:
Description: No serious adverse events were reported, collected, or observed during this study. Total number of participants were 44. Other adverse events were not recorded.
Arm/Group | Normal Saline | Hypertonic Saline
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No